CLINICAL TRIAL: NCT00123474
Title: A Randomized Two-by-Two, Multicenter, Open-Label Phase III Study of BMS-354825 Administered Orally at a Dose of 50 mg or 70 mg Twice Daily or 100 mg or 140 mg Once Daily in Subjects With Chronic Phase Philadelphia Chromosome or BCR-ABL Positive Chronic Myelogenous Leukemia Who Are Resistant or Intolerant to Imatinib Mesylate (Gleevec)
Brief Title: Chronic Myelogenous Leukemia (CML) - Follow on: Study of BMS-354825 in Subjects With CML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-034
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Myeloid Leukemia, Chronic, Chronic-Phase
Keywords: Chronic Phase Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: dasatinib
- 2 (Experimental)
  Interventions: Drug: dasatinib
- 3 (Experimental)
  Interventions: Drug: dasatinib
- 4 (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Tablets, Oral, 50 mg BID, indefinitely, survival study
  Other Names: Sprycel; BMS-354825
  Arms: 1
Drug: dasatinib — Tablets, Oral, 70 mg BID, indefinitely, survival study
  Other Names: Sprycel; BMS-354825
  Arms: 2
Drug: dasatinib — Tablets, Oral, 100 mg QD, indefinitely, survival study
  Other Names: Sprycel; BMS-354825
  Arms: 3
Drug: dasatinib — Tablets, Oral, 140 mg QD, indefinitely, survival study
  Other Names: Sprycel; BMS-354825
  Arms: 4

SUMMARY:
This is a phase III study of BMS-354825 in subjects with chronic phase Philadelphia chromosome or BCR-ABL positive chronic myelogenous leukemia, who are resistant or intolerant to imatinib mesylate (Gleevec).

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Subjects with Philadelphia chromosome positive (Ph+) (or BCR/ABL+) chronic phase chronic myeloid leukemia whose disease has primary or acquired hematologic resistance to imatinib mesylate or who are intolerant of imatinib mesylate.
* Men and women, 18 years or older
* Adequate hepatic function
* Adequate renal function
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month before and at least 3 months after the study in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Subjects who are eligible and willing to undergo transplantation during the screening period
* A serious uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy
* Uncontrolled or significant cardiovascular disease
* Medications that increase bleeding risk
* Medications that change heart rhythms
* Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
* History of significant bleeding disorder unrelated to CML
* Concurrent incurable malignancy other than CML
* Evidence of organ dysfunction or digestive dysfunction that would prevent administration of study therapy
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2005-07; Primary Completion 2006-09 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (134):
- United States (40):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Central Hematology Oncology Medical Group Inc., Alhambra, California
  - Pacific Cancer Medical Center Inc, Anaheim, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - Pacific Shores Medical Group, Long Beach, California
  - Ucla Dept. Of Medicine, Los Angeles, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Georgetown University Med Ctr, Washington D.C., District of Columbia
  - Washington Cancer Institute At Washington Hospital Center, Washington D.C., District of Columbia
  - University Of Florida, Gainesville, Florida
  - University Of Miami, Miami, Florida
  - Md Anderson Cancer Center Orlando, Orlando, Florida
  - Emory University School Of Medicine, Atlanta, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Gwinnett Hospital System Inc., Lawrenceville, Georgia
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - University Of Chicago, Chicago, Illinois
  - Oncology Hematology Associates Of Central Illinois, Pc, Peoria, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University Of Kansas Medical Center, Westwood, Kansas
  - University Of Kentucky, Lexington, Kentucky
  - University Of Maryland, Baltimore, Maryland
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Devetten, Marcel, Omaha, Nebraska
  - Nevada Cancer Institute, Las Vegas, Nevada
  - The Cancer Center At Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute Of New Jersey, New Brunswick, New Jersey
  - New York Presbyterian Hospital, New York, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Ut Southwestern Medical Center, Dallas, Texas
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Argentina (4):
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Buenos Aires
  - Local Institution, Capital Federal
  - Local Institution, Córdoba
- Australia (6):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, St Leonards, New South Wales
  - Local Institution, South Brisbane, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, East Melbourne, Victoria
  - Local Institution, Perth, Western Australia
- Local Institution, Vienna, Austria
- Belgium (6):
  - Local Institution, B-leuven
  - Local Institution, Bruges
  - Local Institution, Brussels
  - Local Institution, Charleroi
  - Local Institution, Edegem
  - Local Institution, Yvoir
- Brazil (5):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, São Paulo, São Paulo
  - Local Institution, CEP - Campinas
  - Local Institution, San Paulo, Sp
- Canada (3):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Hamilton, Ontario
  - Local Institution, Montreal, Quebec
- Czechia (2):
  - Local Institution, Brno
  - Local Institution, Prague
- Denmark (3):
  - Local Institution, Aarhus C
  - Local Institution, Herlev
  - Local Institution, Odense C
- Local Institution, Helsinki, Finland
- France (11):
  - Local Institution, Cedex, Pierre Benite
  - Local Institution, Caen
  - Local Institution, Créteil
  - Local Institution, Grenoble
  - Local Institution, Lille
  - Local Institution, Marseille
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
- Germany (6):
  - Local Institution, Dresden
  - Local Institution, Frankfurt am Main
  - Local Institution, Hamburg
  - Local Institution, Leipzig
  - Local Institution, Mainz
  - Local Institution, Mannheim
- Local Institution, Budapest, Hungary
- Ireland (2):
  - Local Institution, Co Galway, Galway
  - Local Institution, Dublin
- Local Institution, Ramat Gan, Israel
- Italy (5):
  - Local Institution, Bari
  - Local Institution, Monza (mi)
  - Local Institution, Napoli
  - Local Institution, Orbassano
  - Local Institution, Roma
- Local Institution, Distrito Federal, Mexico
- Netherlands (2):
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
- Local Institution, Trondheim, Norway
- Peru (2):
  - Local Institution, Lima, Lima Province
  - Local Institution, Jesus Maria, Lima region
- Local Institution, Quezon City, Philippines
- Poland (6):
  - Local Institution, Gdansk
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Warsaw
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Local Institution, Singapore, Singapore
- South Africa (5):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Groenkloof, Gauteng
  - Local Institution, Parktown, Gauteng
  - Local Institution, Soweto, Gauteng
  - Local Institution, Observatory, Western Cape
- South Korea (3):
  - Local Institution, Jeollanam-do
  - Local Institution, Kyunggi-do
  - Local Institution, Seoul
- Spain (2):
  - Local Institution, Madrid
  - Local Institution, Pamplona
- Sweden (2):
  - Local Institution, Lund
  - Local Institution, Uppsala
- Local Institution, Basel, Switzerland
- Taiwan (2):
  - Local Institution, Taipei
  - Local Institution, Taoyuan
- United Kingdom (6):
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution, London, Greater London
  - Local Institution, Liverpool, Merseyside
  - Local Institution, Newcastle, Tyne and Wear
  - Local Institution, Birmingham, West Midlands
  - Local Institution, Glasgow

REFERENCES:
- [Background] Porkka K, Khoury HJ, Paquette RL, Matloub Y, Sinha R, Cortes JE. Dasatinib 100 mg once daily minimizes the occurrence of pleural effusion in patients with chronic myeloid leukemia in chronic phase and efficacy is unaffected in patients who develop pleural effusion. Cancer. 2010 Jan 15;116(2):377-86. doi: 10.1002/cncr.24734. PMID 19924787
- [Background] Muller MC, Cortes JE, Kim DW, Druker BJ, Erben P, Pasquini R, Branford S, Hughes TP, Radich JP, Ploughman L, Mukhopadhyay J, Hochhaus A. Dasatinib treatment of chronic-phase chronic myeloid leukemia: analysis of responses according to preexisting BCR-ABL mutations. Blood. 2009 Dec 3;114(24):4944-53. doi: 10.1182/blood-2009-04-214221. Epub 2009 Sep 24. PMID 19779040
- [Background] Shah NP, Kantarjian HM, Kim DW, Rea D, Dorlhiac-Llacer PE, Milone JH, Vela-Ojeda J, Silver RT, Khoury HJ, Charbonnier A, Khoroshko N, Paquette RL, Deininger M, Collins RH, Otero I, Hughes T, Bleickardt E, Strauss L, Francis S, Hochhaus A. Intermittent target inhibition with dasatinib 100 mg once daily preserves efficacy and improves tolerability in imatinib-resistant and -intolerant chronic-phase chronic myeloid leukemia. J Clin Oncol. 2008 Jul 1;26(19):3204-12. doi: 10.1200/JCO.2007.14.9260. Epub 2008 Jun 9. PMID 18541900
- [Derived] Shah NP, Rousselot P, Schiffer C, Rea D, Cortes JE, Milone J, Mohamed H, Healey D, Kantarjian H, Hochhaus A, Saglio G. Dasatinib in imatinib-resistant or -intolerant chronic-phase, chronic myeloid leukemia patients: 7-year follow-up of study CA180-034. Am J Hematol. 2016 Sep;91(9):869-74. doi: 10.1002/ajh.24423. Epub 2016 Jun 20. PMID 27192969
- [Derived] Shah NP, Guilhot F, Cortes JE, Schiffer CA, le Coutre P, Brummendorf TH, Kantarjian HM, Hochhaus A, Rousselot P, Mohamed H, Healey D, Cunningham M, Saglio G. Long-term outcome with dasatinib after imatinib failure in chronic-phase chronic myeloid leukemia: follow-up of a phase 3 study. Blood. 2014 Apr 10;123(15):2317-24. doi: 10.1182/blood-2013-10-532341. Epub 2014 Feb 25. PMID 24569263
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated July 2005 and completed July 2014.
Pre-assignment Details: 724 participants were enrolled, 670 were randomized, and 662 were treated with study drug. Reasons for non-randomization: 38 no longer met criteria, 8 other reasons, 7 withdrew consent, and 1 death.
Groups:
- Dasatinib 100 mg QD: Participants received 100 mg once a day (QD) until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
- Dasatinib 140 mg QD: Participants received 140 mg QD until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
- Dasatinib 50 mg BID: Participants received 50 mg twice a day (BID) until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw. After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing schedule were allowed to switch to a QD dosing schedule.
- Dasatinib 70 mg BID: Participants received 70 mg BID until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw. After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing schedule were allowed to switch to a QD dosing schedule.
Period: Randomized to Treatment
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Started | 167 | 167 | 168 | 168
Completed | 166 | 163 | 166 | 167
Not Completed | 1 | 4 | 2 | 1
Not completed — Randomized, never treated | 1 | 4 | 2 | 1
Period: As Treated at Study Closure
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Started | 165 (Randomized to 50 mg BID but received 100 mg QD.) | 163 | 167 | 167
Completed | 0 | 0 | 0 (Randomized to 100 mg QD but received 50 mg BID.) | 0
Not Completed | 165 | 163 | 167 | 167
Not completed — not reported when site closed | 1 | 0 | 1 | 0
Not completed — Adverse Event | 10 | 4 | 10 | 8
Not completed — Disease Progression | 35 | 42 | 29 | 27
Not completed — Investigator Request | 12 | 6 | 7 | 5
Not completed — non-specified | 54 | 47 | 57 | 60
Not completed — Study Drug Toxicity | 39 | 45 | 45 | 51
Not completed — Withdrawal by Subject | 14 | 19 | 18 | 16

BASELINE CHARACTERISTICS:
Population: All participants randomized to a treatment arm are summarized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID | Total
Number analyzed (Participants) | 167 | 167 | 168 | 168 | 670
Age, Customized [Number; unit: participants]
  Less than, equal to (<=) 65 years | 121 | 128 | 130 | 125 | 504
  Greater than (>) 65 years | 46 | 39 | 38 | 43 | 166
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 97 | 83 | 91 | 354
  Male | 84 | 70 | 85 | 77 | 316
Imatinib Status [Number; unit: participants] — Primary Resistance: no decrease in white blood cell (WBC) count after ≥ 4 weeks imatinib or not achieved a complete hematologic response (CHR) after 3 months, a major cytogenetic response (MCyR) after 6 months, or a complete cytogenetic response (CCyR) after 12 months. Acquired resistance: achieved MCyR and no longer met the criteria for MCyR. Intolerance: Grade ≥ 3 toxicity considered at least possibly related to imatinib at a dose of ≤ 400 mg/day which led to discontinuation of therapy; tolerated the dose of 400 mg but did not achieve a CCyR and subsequently did not tolerate doses ≥ 600 mg.
  participants
    Primary Resistance to Imatinib | 75 | 78 | 88 | 81 | 322
    Acquired Resistance to Imatinib | 49 | 45 | 36 | 45 | 175
    Intolerant to Imatinib | 43 | 44 | 44 | 42 | 173

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Major Cytogenetic Response (MCyR) at 6 Months Follow-Up
Description: Cytogenetic response (CyR) was based on the number of Philadelphia chromosome positive (Ph+) metaphases among cells in metaphase on a Bone Marrow (BM) sample. The criteria for CyR were as follows: Complete cytogenetic response (CCyR): 0% Ph+ cells in metaphase in BM; Partial cytogenetic response (PCyR): >0 to 35% Ph+ cells in metaphase in BM; Minor cytogenetic response: >35 to 65% Ph+ cells in metaphase in BM; Minimal cytogenetic response: >65 to 95% Ph+ cells in metaphase in BM; No cytogenetic response: >95 to 100% Ph+ cells in metaphase in BM; Best CyR was defined as the best response obtained at any time during the study; MCyR was defined as a best CyR of complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR). Baseline=closest to, but no later than, the first day of study drug for treated participants and closest to, but no later than, the date of randomization, for those who were randomized but who never received treatment, unless otherwise specified.
Time Frame: 6 months
Population: All randomized imatinib-resistant participants with available data were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Groups:
- QD Dasatinib: Participants received either 100 mg or 140 mg once a day (QD) dasatinib until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
- BID Dasatinib: Participants received either 50 mg or 70 mg twice a day (BID) dasatinib until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
Arm/Group | QD Dasatinib | BID Dasatinib
Number analyzed (Participants) | 247 | 251
percentage of Participants | 51.8 [45.4 to 58.2] | 49.0 [42.7 to 55.4]
Statistical Analysis 1: Comparison: QD Dasatinib vs BID Dasatinib; 6 Month Analysis; Test type: Non-Inferiority or Equivalence — Non-inferiority of the QD schedule relative to the BID schedule was deduced if the lower bound of the 95% confidence interval (CI) for the MCyRRQD minus MCyRRBID difference was greater than or equal to -15%; Risk Difference (RD) = 2.8, 95% CI 2-sided [-6.0 to 11.6]

2. Secondary Outcome: Percent of Participants With MCyR At or Prior to 24 Months Follow-Up
Description: CyR was based on the number of Ph+ metaphases among cells in metaphase on a Bone Marrow (BM) sample. The criteria for CyR were as follows: CCyR: 0% Ph+ cells in metaphase in BM; PCyR: >0 to 35% Ph+ cells in metaphase in BM; Minor cytogenetic response: >35 to 65% Ph+ cells in metaphase in BM; Minimal cytogenetic response: >65 to 95% Ph+ cells in metaphase in BM; No cytogenetic response: >95 to 100% Ph+ cells in metaphase in BM; Best CyR was defined as the best response obtained at any time during the study; MCyR was defined as a best CyR of CCyR or PCyR. Baseline=closest to, but no later than, the first day of study drug for treated participants and closest to, but no later than, the date of randomization, for those who were randomized but who never received treatment, unless otherwise specified.
Time Frame: 24 months
Population: All randomized imatinib-resistant participants with available data were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Groups:
- Dasatinib QD: Participants received either 100 mg QD or 140 mg QD until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
- Dasatinib BID: Participants received either 50 mg BID or 70 mg BID until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw. After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing schedule were allowed to switch to a QD dosing schedule.
- Dasatinib 100 mg Total Daily Dose: Participants received 100 mg as a total daily dose (either 50 mg BID or 100 mg QD) until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
- Dasatinib 140 mg Total Daily Dose: Participants received 140 mg as a total daily dose (either 70 mg BID or 140 mg QD) until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
Arm/Group | Dasatinib QD | Dasatinib BID | Dasatinib 100 mg Total Daily Dose | Dasatinib 140 mg Total Daily Dose
Number analyzed (Participants) | 247 | 250 | 248 | 249
percentage of Participants | 58.3 [51.9 to 64.5] | 56.4 [50.0 to 62.6] | 57.3 [50.8 to 63.5] | 57.4 [51.0 to 63.7]
Statistical Analysis 1: Comparison: Dasatinib QD vs Dasatinib BID; Test type: Non-Inferiority or Equivalence — Non-inferiority of the QD schedule relative to the BID schedule was deduced if the lower bound of the 95% CI for the MCyRRQD minus MCyRRBID difference was greater than or equal to -15%; Risk Difference (RD) = 1.9, 95% CI 2-sided [-6.8 to 10.6]
Statistical Analysis 2: Comparison: Dasatinib 100 mg Total Daily Dose vs Dasatinib 140 mg Total Daily Dose; Test type: Non-Inferiority or Equivalence — Non-inferiority of 100 mg total daily dose relative to 140 mg total daily dose was deduced if the lower bound of the 95% CI for the difference was greater than or equal to -15%; Risk Difference (RD) = -0.2, 95% CI 2-sided [-8.9 to 8.5]

3. Secondary Outcome: Percent of Participants With Complete Hematologic Response (CHR) at 6 and 24 Months Follow-Up
Description: A complete hematologic response (CHR) was obtained when all the following criteria were met: White Blood Cells (WBC) ≤ institutional upper limit of normal (ULN); Platelets < 450,000/mm³; No blasts or promyelocytes in peripheral blood (PB); < 5% myelocytes plus metamyelocytes in PB; Basophils in PB < 20%; No extramedullary involvement (including no splenomegaly or hepatomegaly). Hematologic responses were counted anytime following 14 days after the dosing start date.
Time Frame: 6 months, 24 months
Population: All randomized imatinib-resistant participants with available data were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dasatinib 100 mg QD: Participants received 100 mg QD until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
  After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing schedule were allowed to switch to a QD dosing schedule.
- Dasatinib 140 mg QD: Participants received 140 mg QD until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw. After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing schedule were allowed to switch to a QD dosing schedule.
- Dasatinib 50 mg BID: Participants received 50 mg BID until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw. After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing schedule were allowed to switch to a QD dosing schedule.
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 124 | 123 | 124 | 127
percentage of participants
  6 Months (n=124,123,124,127) | 86.3 [79.0 to 91.8] | 85.4 [77.9 to 91.1] | 91.1 [84.7 to 95.5] | 87.4 [80.3 to 92.6]
  24 Month (n=124,123,124,126) | 88.7 [81.8 to 93.7] | 86.2 [78.8 to 91.7] | 91.9 [85.7 to 96.1] | 88.9 [82.1 to 93.8]

4. Secondary Outcome: Time to MCyR in Participants With MCyR at 6 Months Follow-Up
Description: Time to MCyR was defined as the time from the first dosing date until criteria were first met for CCyR or PCyR, whichever occurred first. Non-responders were censored at the maximum time of all participants in their respective group (ie, maximum between time to MCyR response for responders and time to last cytogenetic assessment for non-responders).
Time Frame: 6 months
Population: Randomized imatinib-resistant participants with MCyR and available data were summarized.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Dasatinib 100 mg QD: Participants received 100 mg once a day (QD) until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
  After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing schedule were allowed to switch to a QD dosing schedule.
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 66 | 62 | 58 | 65
Months | 2.8 [2.8 to 3.0] | 2.8 [2.8 to 2.9] | 2.8 [2.8 to 2.9] | 2.8 [2.8 to 3.0]

5. Secondary Outcome: Time to CHR in Participants With CHR at 6 Months Follow-Up
Description: Time to CHR was defined as the time from the first dosing date until criteria are first met for the response. Non-responders were censored at the maximum time of all participants in their respective group (ie, maximum between time to CHR response for responders and time to last hematologic assessment for non-responders).
Time Frame: 6 months
Population: Randomized imatinib-resistant participants with CHR and available data were summarized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 107 | 105 | 113 | 111
Months | 0.5 [0.5 to 0.6] | 0.5 [0.5 to 0.7] | 0.6 [0.6 to 0.9] | 0.7 [0.5 to 0.9]

6. Secondary Outcome: Time to MCyR in Participants With MCyR at 24 Months Follow-Up
Description: Time to MCyR was defined as the time from the first dosing date until criteria were first met for CCyR or PCyR, whichever occurred first. Non-responders were censored at the maximum time of all participants in their respective group (ie, maximum between time to MCyR response for responders and time to last cytogenetic assessment for non-responders). Cytogenetic assessments were not done after the 2 Year Follow-up.
Time Frame: 24 months
Population: Randomized imatinib-resistant participants with MCyR were summarized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 73 | 71 | 69 | 72
Months | 2.9 [2.8 to 3.4] | 2.8 [2.8 to 3.0] | 2.9 [2.8 to 3.3] | 2.9 [2.8 to 3.0]

7. Secondary Outcome: Time to CHR in Participants With CHR At 24 Months Follow-Up
Description: Time to CHR was defined as the time from the first dosing date until criteria are first met for the response. Non-responders were censored at the maximum time of all participants in their respective group (ie, maximum between time to CHR response for responders and time to last hematologic assessment for non-responders). Cytogenetic assessments were not done after the 2 Year Follow-up.
Time Frame: 24 months
Population: Randomized imatinib-resistant participants with CHR were summarized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 110 | 106 | 114 | 112
Months | 0.5 [0.5 to 0.6] | 0.5 [0.5 to 0.7] | 0.6 [0.5 to 0.9] | 0.7 [0.5 to 0.9]

8. Secondary Outcome: Number of Participants With MCyR Whose Disease Progressed by 24 Months
Description: Progression in a participant=participant achieved a CHR and no longer met the criteria consistently over consecutive 2-weeks after starting their maximum dose; had no CHR after receiving their maximum dose and had an increase in white blood count (WBC) defined as a doubling of the count from the lowest value to >20,000/mm^3 or an increase by > 50,000/mm^3 on two assessments performed at least 2 weeks apart; participant met criteria of accelerated or blast phase CML at any time; had a MCyR and subsequently no longer met the criteria for MCyR after starting their maximum dose; had a ≥ 30% absolute increase in the number of Ph+ metaphases. Although a related secondary endpoint was estimated duration of MCyR, medium duration of MCyR could not be estimated because the majority of participants with MCyR continued to respond, or could not be reliably estimated because of the large number of censored participants. Cytogenetic assessments were not done after the 24 month follow-up.
Time Frame: 24 months
Population: All imatinib-resistant participants who had achieved MCyR and experienced disease progression were summarized.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 73 | 71 | 69 | 72
participants | 5 | 17 | 6 | 9

9. Secondary Outcome: Number of Participants With CHR Whose Disease Progressed by 24 Months
Description: Progression in a participant=achieved a CHR and subsequently no longer met the criteria consistently over a consecutive 2-week period after starting their maximum dose; had no CHR after receiving their maximum dose and had an increase in white blood count (WBC) defined as a doubling of the count from the lowest value to >20,000/mm^3 or an increase by > 50,000/mm^3 on two assessments performed at least 2 weeks apart; met the criteria of accelerated or blast phase CML at any time; had a MCyR and subsequently no longer met the criteria for MCyR after starting their maximum dose; had a ≥ 30% absolute increase in the number of Ph+ metaphases. Although a related secondary endpoint was estimated duration of CHR, medium duration of CHR could not be estimated because the majority of participants with CHR continued to respond, or could not be reliably estimated because of the large number of censored participants.
Time Frame: 24 months
Population: All imatinib-resistant participants who achieved CHR and then experienced disease progression were summarized.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 110 | 106 | 114 | 112
participants | 18 | 28 | 22 | 24

10. Secondary Outcome: Number of Participants With MCyR and Baseline BCR-ABL Gene Mutation - All Treated Participants
Description: BCR-ABL mutations were assessed in participants prior to the start of study drug (baseline) and at the time of disease progression or at end of therapy. Quantification of BCR-ABL transcripts in peripheral blood was evaluated using quantitative reverse transcriptase polymerase chain reaction (Q-RT-PCR, RT-PCR).
Time Frame: Baseline up to 24 months
Population: All randomized, treated participants with available mutation data were summarized.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 147 | 139 | 149 | 146
participants
  Imatinib-resistant Mutations | 49 | 49 | 62 | 48
  Mutations with unknown Imatinib-resistance status | 0 | 1 | 1 | 2
  Imatinib Resistant or unknown mutations | 49 | 50 | 63 | 50
  Polymorphisms | 0 | 2 | 0 | 0
  No Mutations | 98 | 87 | 86 | 96

11. Secondary Outcome: Percent of Imatinib-Resistant Participants With Progression Free Survival (PFS) at 24, 36, 48, 60, 72, and 84 Months Follow-Up
Description: PFS= time from randomization until: CHR achieved and participant subsequently no longer met criteria for CHR over 2 weeks; no CHR after receiving maximum dose and an increase in WBC (ie, doubling of the count from the lowest value to > 20,000/mm^3 or an increase by > 50,000/mm^3 on 2 assessments performed 2 weeks apart); participant met criteria of accelerated phase or blast phase CML; participant had MCyR and subsequently no longer met criteria for MCyR after starting maximum dose; participant had a ≥ 30% absolute increase in number of Ph+ metaphases. Deaths without a reported prior progression were considered to have progressed on the date of death; those who neither progressed nor died were censored on the date of their last cytogenetic or hematologic assessment. When first progression reported during follow-up, it was censored at last on-study assessment. If the first progression reported during follow-up was death, participant considered to have progressed at date of death.
Time Frame: 24, 36, 48, 60, 72, and 84 months
Population: All randomized imatinib-resistant participants were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 124 | 123 | 124 | 126
percentage of participants
  24 Months (n=124,123,124, 127) | 75.2 [66.3 to 82.1] | 61.3 [52.7 to 69.6] | 70.3 [60.8 to 77.9] | 70.8 [61.6 to 78.2]
  36 Months (n=124,123,124, 127) | 64.8 [55.2 to 72.9] | 47.4 [37.7 to 56.5] | 67.1 [57.3 to 75.1] | 58.2 [48.4 to 66.8]
  48 Months (n=124,123,124, 127) | 57.8 [48.0 to 66.5] | 40.0 [30.6 to 49.3] | 63.8 [53.7 to 72.2] | 55.1 [45.2 to 64.8]
  60 Months (n=124,123,124, 127) | 50.2 [40.2 to 59.3] | 36.4 [27.1 to 45.8] | 57.4 [46.9 to 66.5] | 50.2 [40.2 to 59.4]
  72 Months (n=124,123,124, 127) | 44.0 [34.0 to 53.6] | 31.4 [22.4 to 40.8] | 50.7 [40.0 to 60.4] | 45.3 [35.2 to 54.8]
  84 Months (n=124,123,124, 127) | 39.0 [29.2 to 48.7] | 30.2 [21.2 to 39.6] | 42.1 [31.5 to 52.4] | 41.3 [31.3 to 51.0]

12. Secondary Outcome: Percent of Imatinib-Resistant Participants With Overall Survival (OS) at 24, 36, 48, 60, 72, and 84 Months Follow-Up
Description: Overall survival (OS) was defined as the time from randomization until death. Survival data were collected for up to 5 years on participants who had discontinued dasatinib treatment. Participants who did not die or who were lost to follow-up were censored on the last date the participant was known to be alive.
Time Frame: 24, 36, 48, 60, 72, and 84 months
Population: All randomized imatinib-resistant participants were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 124 | 123 | 124 | 126
percentage of participants
  24 Months (n=124,123,124,127) | 90.1 [83.2 to 94.2] | 93.9 [87.6 to 97.0] | 88.9 [81.6 to 93.4] | 85.1 [77.3 to 90.3]
  36 Months (n=124,123,124,127) | 87.5 [80.2 to 92.3] | 83.8 [75.6 to 89.5] | 83.5 [75.3 to 89.1] | 76.5 [67.7 to 83.1]
  48 Months (n=124,123,124,127) | 79.7 [71.3 to 85.9] | 82.0 [73.4 to 88.0] | 80.7 [72.1 to 86.9] | 71.1 [61.9 to 78.4]
  60 Months (n=124,123,124,127) | 75.1 [66.1 to 82.0] | 78.0 [68.9 to 84.7] | 73.6 [64.1 to 80.9] | 69.1 [59.8 to 76.7]
  72 Months (n=124,123,124,127) | 67.9 [58.3 to 75.8] | 72.6 [62.9 to 80.1] | 71.4 [61.8 to 79.0] | 67.1 [57.6 to 74.9]
  84 Months (n=124,123,124,127) | 62.6 [52.6 to 71.0] | 68.1 [58.0 to 76.2] | 67.9 [57.9 to 76.0] | 65.0 [55.3 to 73.0]

13. Secondary Outcome: Percent of Participants Intolerant to Imatinib With MCyR at 6 Months and at 24 Months Follow-Up, by QD and BID Schedules and by Total Daily Dose
Description: CyR was based on the number of Ph+ metaphases among cells in metaphase on a BM sample. The criteria for CyR were as follows: complete cytogenetic response (CCyR): 0% Ph+ cells in metaphase in BM; PCyR: >0 to 35% Ph+ cells in metaphase in BM; Minor cytogenetic response: >35 to 65% Ph+ cells in metaphase in BM; Minimal cytogenetic response: >65 to 95% Ph+ cells in metaphase in BM; No cytogenetic response: >95 to 100% Ph+ cells in metaphase in BM; Best CyR was defined as the best response obtained at any time during the study; MCyR was defined as a best CyR of CCyR or PCyR.
Time Frame: 6 months, 24 months
Population: All randomized imatinib-intolerant participants with available data were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- QD Dasatinib: Participants received either 100 mg or 140 mg once a day (QD) until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
- BID Dasatinib: Participants received either 50 mg or 70 mg twice a day (BID) until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
- Total Daily Dose 100 mg: Participants received either 100 mg QD or 50 mg BID until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
- Total Daily Dose 140 mg: Participants received either 140 mg QD or 70 mg BID until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
Arm/Group | QD Dasatinib | BID Dasatinib | Total Daily Dose 100 mg | Total Daily Dose 140 mg
Number analyzed (Participants) | 87 | 85 | 87 | 86
percentage of participants
  6 Month | 72.4 [61.8 to 81.5] | 70.6 [59.7 to 80.0] | 73.6 [63.0 to 82.4] | 69.4 [58.5 to 79.0]
  24 Month | 77.0 [66.8 to 85.4] | 75.6 [65.1 to 84.2] | 77.0 [66.8 to 85.4] | 75.6 [65.1 to 84.2]
Statistical Analysis 1: Comparison: QD Dasatinib vs BID Dasatinib; 6 Month Analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Risk Difference (RD) = 1.8, 95% CI 2-sided [-11.7 to 15.3]
Statistical Analysis 2: Comparison: Total Daily Dose 100 mg vs Total Daily Dose 140 mg; 6 Month Analysis; Test type: Non-Inferiority or Equivalence — Non-inferiority of 100 mg QD Total Daily Dose relative to 140 mg QD Total Daily Dose was deduced if the lower bound of the 95% CI difference was greater than or equal to -15%; Risk Difference (RD) = 4.2, 95% CI 2-sided [-9.3 to 17.6]
Statistical Analysis 3: Comparison: QD Dasatinib vs BID Dasatinib; 24 Month Analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Risk Difference (RD) = 1.4, 95% CI 2-sided [-11.2 to 14.1]
Statistical Analysis 4: Comparison: Total Daily Dose 100 mg vs Total Daily Dose 140 mg; 24 Month Analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 2]; Risk Difference (RD) = 1.4, 95% CI 2-sided [-11.2 to 14.1]

14. Secondary Outcome: Percent of Participants Intolerant to Imatinib With CHR at 6 Months and at 24 Months Follow-Up
Description: A CHR was obtained when all the following criteria were met: White Blood Cells (WBC) ≤ institutional upper limit of normal (ULN); Platelets < 450,000/mm³; No blasts or promyelocytes in peripheral blood (PB); < 5% myelocytes plus metamyelocytes in PB; Basophils in PB < 20%; No extramedullary involvement (including no splenomegaly or hepatomegaly). Hematologic responses were counted anytime following 14 days after the dosing start date.
Time Frame: 6 months, 24 months
Population: All randomized imatinib-intolerant participants were summarized.
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 43 | 44 | 44 | 42
percentage of participants
  6 Months (n=43,44,44,41) | 100 | 86 | 93 | 85
  24 Months (n=43,44,44,42) | 100 | 89 | 93 | 86

15. Secondary Outcome: Percent of Imatinib Intolerant Participants With Progression Free Survival After 24, 36, 48, 60, 72, and 84 Months of Follow-Up
Description: as for outcome 11
Time Frame: 24, 36, 48, 60, 72, and 84 months
Population: All randomized imatinib-intolerant participants with available data were summarized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 100mg QD: Participants received 100 mg QD until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
  After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing schedule were allowed to switch to a QD dosing schedule.
- 140mg QD: Participants received 140 mg QD until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw. After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing.
- 50mg BID: Participants received 50 mg BID until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw. After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing.
- 70mg BID: Participants received 70 mg BID until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw. After the 2-year analysis, and with Protocol Amendment 02, participants on a BID dosing.
Arm/Group | 100mg QD | 140mg QD | 50mg BID | 70mg BID
Number analyzed (Participants) | 43 | 44 | 44 | 42
percentage of participants
  24 Months (n=43,44,44,42) | 83.6 [67.0 to 92.3] | 87.7 [72.8 to 94.7] | 77.4 [61.0 to 87.6] | 83.7 [67.1 to 92.4]
  36 Months (n=43,44,44,42) | 71.7 [53.6 to 83.7] | 76.0 [58.7 to 86.8] | 68.6 [51.1 to 80.9] | 77.4 [59.6 to 88.1]
  48 Months (n=43,44,44,42) | 62.7 [44.5 to 76.5] | 76.0 [58.7 to 86.8] | 62.0 [44.1 to 75.7] | 66.9 [47.8 to 80.4]
  60 Months (n=43,44,44,42) | 59.2 [40.8 to 73.6] | 71.2 [52.1 to 83.8] | 62.0 [44.1 to 75.7] | 59.5 [40.1 to 74.4]
  72 Months (n=43,44,44,42) | 59.2 [40.8 to 73.6] | 66.5 [46.3 to 80.6] | 58.2 [39.8 to 72.7] | 55.2 [35.7 to 71.1]
  84 Months (n=43,44,44,42) | 50.9 [32.1 to 67.0] | 66.5 [46.3 to 80.6] | 47.5 [27.4 to 65.2] | 50.2 [30.4 to 67.1]

16. Secondary Outcome: Percent of Imatinib Intolerant Participants With Overall Survival After 24, 36, 48, 60, 72, and 84 Months of Follow-up
Description: as for outcome 12
Time Frame: 24, 36, 48, 60, 72, and 84 months
Population: All randomized imatinib-intolerant participants were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mg QD | 140mg QD | 50mg BID | 70mg BID
Number analyzed (Participants) | 43 | 44 | 44 | 42
percentage of participants
  24 Months (n=43,44,44,42) | 94.9 [81.2 to 98.7] | 92.8 [79.2 to 97.6] | 95.3 [82.5 to 98.8] | 97.4 [82.8 to 99.6]
  36 Months (n=43,44,44,42) | 89.7 [74.9 to 96.0] | 92.8 [79.2 to 97.6] | 90.4 [76.4 to 96.3] | 94.7 [80.6 to 98.7]
  48 Months (n=43,44,44,42) | 84.5 [68.6 to 92.7] | 87.5 [72.4 to 94.6] | 85.1 [69.7 to 93.0] | 86.8 [71.2 to 94.3]
  60 Months (n=43,44,44,42) | 81.8 [65.6 to 90.9] | 87.5 [72.4 to 94.6] | 82.4 [66.6 to 91.2] | 81.1 [64.3 to 90.5]
  72 Months (n=43,44,44,42) | 79.0 [62.3 to 88.9] | 87.5 [72.4 to 94.6] | 79.6 [63.2 to 89.3] | 81.1 [64.3 to 90.5]
  84 Months (n=43,44,44,42) | 70.0 [52.2 to 82.2] | 87.5 [72.4 to 94.6] | 76.6 [59.7 to 87.2] | 77.7 [60.1 to 88.2]

17. Secondary Outcome: Percent of All Randomized Participants With Cytogenic and Hematologic Response by Dosing Schedule (QD or BID) and by Total Daily Dose (100 mg or 140 mg) at 6 Months Follow-Up
Description: Complete cytogenetic response (CCyR): 0% Ph+ cells in metaphase in BM. Partial cytogenetic response (PCyR): >0 to 35% Ph+ cells in metaphase in BM. MCyR: best cytogenetic response of CCyR or PCyR. A complete hematologic response (CHR) was obtained when all the following criteria were met: White Blood Cells (WBC) ≤ institutional upper limit of normal (ULN); Platelets < 450,000/mm³; No blasts or promyelocytes in peripheral blood (PB); < 5% myelocytes plus metamyelocytes in PB; Basophils in PB < 20%; No extramedullary involvement (including no splenomegaly or hepatomegaly). Hematologic responses were counted anytime following 14 days after the dosing start date.
Time Frame: 6 months
Population: All randomized participants were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QD Dasatinib | BID Dasatinib | Total Daily Dose 100 mg | Total Daily Dose 140 mg
Number analyzed (Participants) | 334 | 336 | 335 | 335
percentage of participants
  MCyR (n=334,336,335,335) | 57.2 [51.7 to 62.6] | 54.5 [49.0 to 59.9] | 56.1 [50.6 to 61.5] | 55.5 [50.0 to 60.9]
  CHR(n=334,336,335,335) | 87.7 [83.7 to 91.0] | 89.3 [85.5 to 92.4] | 90.7 [87.1 to 93.6] | 86.3 [82.1 to 89.8]

18. Secondary Outcome: Percent of All Randomized Participants With Cytogenic and Hematologic Response by Dosing Schedule (QD or BID) and by Total Daily Dose (100 mg or 140 mg) at 24 Months Follow-Up
Description: Complete cytogenetic response (CCyR): 0% Ph+ cells in metaphase in BM. Partial cytogenetic response (PCyR): >0 to 35% Ph+ cells in metaphase in BM. MCyR: best cytogenetic response of CCyR or PCyR. A complete hematologic response (CHR) was obtained when all the following criteria were met: White Blood Cells (WBC) ≤ institutional upper limit of normal (ULN); Platelets < 450,000/mm³; No blasts or promyelocytes in peripheral blood (PB); < 5% myelocytes plus metamyelocytes in PB; Basophils in PB < 20%; No extramedullary involvement (including no splenomegaly or hepatomegaly). Hematologic responses were counted anytime following 14 days after the dosing start date. No cytogenic assessments were made after 2 years of follow-up.
Time Frame: 24 months
Population: All randomized participants were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | QD Dasatinib | BID Dasatinib | Total Daily Dose 100 mg | Total Daily Dose 140 mg
Number analyzed (Participants) | 334 | 336 | 335 | 335
percentage of participants
  MCyR(n=334,336,335,335) | 63.2 [57.8 to 68.4] | 61.3 [55.9 to 66.5] | 62.4 [57.0 to 67.6] | 62.1 [56.7 to 67.3]
  CHR (n=334,336,335,335) | 89.2 [85.4 to 92.3] | 90.2 [86.5 to 93.1] | 91.9 [88.5 to 94.6] | 87.5 [83.4 to 90.8]

19. Secondary Outcome: Percent of Participants With Progression Free Survival (PFS) at 24, 36, 48, 60, 72, and 84 Months Follow-Up by Dose Schedule and Total Daily Dose - All Randomized Participants
Description: as for outcome 11
Time Frame: 24, 36, 48, 60, 72, and 84 months
Population: All participants who were randomized to a treatment arm were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 167 | 167 | 168 | 168
percentage of participants
  24 Months (n=167, 167, 168, 168) | 77.4 [69.9 to 83.2] | 67.7 [59.6 to 74.5] | 72.2 [64.3 to 78.7] | 73.9 [66.1 to 80.1]
  36 Months (n=167, 167, 168, 168) | 66.6 [58.3 to 73.6] | 54.0 [45.4 to 61.8] | 67.5 [59.2 to 74.5] | 62.8 [54.3 to 70.1]
  48 Months (n=167, 167, 168, 168) | 59.1 [50.6 to 66.6] | 48.0 [39.4 to 56.2] | 63.3 [54.8 to 70.7] | 58.7 [50.1 to 66.3]
  60 Months (n=167, 167, 168, 168) | 52.5 [43.8 to 60.5] | 44.2 [35.5 to 52.5] | 58.7 [49.8 to 66.5] | 52.5 [43.7 to 60.5]
  72 Months (n=167, 167, 168, 168) | 40.0 [39.2 to 56.2] | 39.2 [30.6 to 47.7] | 52.8 [43.7 to 61.1] | 47.7 [38.7 to 56.0]
  84 Months (n=167, 167, 168, 168) | 42.1 [33.4 to 50.6] | 38.2 [29.6 to 46.7] | 43.9 [34.5 to 52.9] | 43.5 [34.5 to 52.1]

20. Secondary Outcome: Percent of Participants Overall Survival at 24, 36, 48, 60, 72, and 84 Months Follow-Up - All Randomized Participants
Description: as for outcome 12
Time Frame: 24, 36, 48, 60, 72, and 84 months
Population: All participants who were randomized to a treatment arm were summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 167 | 167 | 168 | 168
percentage of participants
  24 Months (n=167, 167, 168, 168) | 91.3 [85.8 to 94.8] | 93.6 [88.4 to 96.5] | 90.6 [84.9 to 94.2] | 88.1 [81.9 to 92.2]
  36 Months (n=167, 167, 168, 168) | 88.1 [82.0 to 92.3] | 86.2 [79.6 to 90.8] | 85.3 [78.7 to 90.0] | 80.9 [73.9 to 86.3]
  48 Months (n=167, 167, 168, 168) | 81.0 [73.9 to 86.3] | 83.4 [76.4 to 88.5] | 81.8 [74.7 to 87.1] | 74.9 [67.3 to 81.0]
  60 Months (n=167, 167, 168, 168) | 76.8 [69.4 to 82.7] | 80.5 [73.1 to 86.0] | 75.9 [68.2 to 82.0] | 72.0 [64.1 to 78.4]
  72 Months (n=167, 167, 168, 168) | 70.9 [62.9 to 77.5] | 76.6 [68.7 to 82.7] | 73.6 [65.6 to 80.0] | 70.5 [62.5 to 77.1]
  84 Months (n=167, 167, 168, 168) | 64.6 [56.1 to 71.8] | 73.4 [65.2 to 79.9] | 70.3 [62.0 to 77.1] | 68.1 [59.8 to 74.9]

21. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Adverse Events (AEs) That Led to Treatment Discontinuation at 24 Months of Follow-up
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Baseline=closest to, but no later than, the first day of study drug for treated participants.
Time Frame: Baseline to 30 days post last dose, up to 24 months
Population: All randomized participants who received at least one dose of study drug were summarized.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg QD | Dasatinib 140 mg QD | Dasatinib 50 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 165 | 163 | 167 | 167
participants
  Any SAE | 58 | 67 | 73 | 78
  Drug-Related SAE | 32 | 40 | 47 | 55
  Drug-Related AEs that led to discontinuationt | 14 | 24 | 20 | 25
  Death within 30 days of last dose | 3 | 2 | 6 | 5

22. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Adverse Events (AEs) That Led toTreatment Discontinuation After 7 Year Follow-up
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Baseline=closest to, but no later than, the first day of study drug for treated participants. After the 2-year analysis and Protocol Amendment 02, those on a BID dosing schedule were allowed to switch to a QD dosing schedule. Due to the large number of participants switching from BID dosing to QD dosing, the abbreviated dosing data collection method incorporated in Amendment 03, the overall safety data are presented for the 100 mg QD group and combined for the other treatment groups.
Time Frame: Baseline to 30 days post last dose, up to 7 years (study closure July 2014)
Population: All randomized participants who received at least one dose of study drug were summarized.
Measure: Number; unit: participants
Groups:
- 100 mg QD: Participants received 100 mg once a day (QD) until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
- Other Treatment Groups: Participants participated in all other treatment arms until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
- Total: Participants received study drug in any schedule or total daily dose until progression of disease, development of intolerable toxicity, or the participant's decision to withdraw.
Arm/Group | 100 mg QD | Other Treatment Groups | Total
Number analyzed (Participants) | 165 | 497 | 662
participants
  All Deaths | 51 | 133 | 184
  Deaths on-study or within 30 days post dose | 11 | 15 | 26
  SAEs | 75 | 259 | 334
  AEs Leading to Discontinuation of Treatment | 43 | 153 | 196

ADVERSE EVENTS:
Time Frame: Baseline to 30 days post last dose, up to 7 years (study closure July 2014)
Arm/Group | 100mg QD | 140mg QD | 50mg BID | 70mg BID
Serious Adverse Events (participants affected / at risk) | 75/165 | 78/163 | 89/167 | 92/167
Other Adverse Events (participants affected / at risk) | 160/165 | 155/163 | 160/167 | 165/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100mg QD (N=165) | 140mg QD (N=163) | 50mg BID (N=167) | 70mg BID (N=167)
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 4 | 3
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 3 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Lung infection (Infections and infestations) | 3 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 | 27 | 18 | 25
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Amaurosis (Eye disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chronic myeloid leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
Infection (Infections and infestations) | 5 | 0 | 2 | 2
Loose tooth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 2 | 2 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 1 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Skin cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 1 | 1
Sudden death (General disorders) | 1 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 5
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anaphylactoid reaction (Immune system disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 4 | 2 | 3 | 3
Clostridium test positive (Investigations) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Device failure (General disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 2 | 2 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4 | 6 | 9
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 1
Blast cell count increased (Investigations) | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 12 | 5 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 8 | 10
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 2 | 3 | 3 | 3
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 3 | 2 | 5
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 1 | 0 | 1
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 2 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2 | 0
Infectious colitis (Infections and infestations) | 0 | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 5 | 6 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Blast cell proliferation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Haemoglobin (Investigations) | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 3
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Thrombosis in device (General disorders) | 0 | 0 | 1 | 0
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 5 | 2 | 0 | 4
Central nervous system haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 2 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 15 | 10 | 8
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 3
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Serositis (General disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 4 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 3 | 1 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Death (General disorders) | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Endocarditis enterococcal (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 1 | 2
Gastroenteritis clostridial (Infections and infestations) | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Medical device pain (General disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 2
Pyrexia (General disorders) | 3 | 11 | 6 | 9
Sepsis (Infections and infestations) | 1 | 1 | 3 | 4
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100mg QD (N=165) | 140mg QD (N=163) | 50mg BID (N=167) | 70mg BID (N=167)
Acne (Skin and subcutaneous tissue disorders) | 5 | 7 | 7 | 9
Hypertension (Vascular disorders) | 15 | 12 | 13 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 | 29 | 24 | 22
Palpitations (Cardiac disorders) | 13 | 7 | 8 | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 41 | 51 | 54 | 51
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 29 | 28 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 53 | 42 | 57 | 54
Erythema (Skin and subcutaneous tissue disorders) | 5 | 7 | 9 | 5
Fatigue (General disorders) | 62 | 62 | 56 | 49
Infection (Infections and infestations) | 9 | 4 | 8 | 2
Nasopharyngitis (Infections and infestations) | 23 | 13 | 22 | 13
Oral herpes (Infections and infestations) | 13 | 5 | 9 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 22 | 17 | 23
Sinusitis (Infections and infestations) | 19 | 8 | 17 | 12
Anaemia (Blood and lymphatic system disorders) | 23 | 14 | 26 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 | 39 | 36 | 30
Chest pain (General disorders) | 21 | 16 | 19 | 17
Constipation (Gastrointestinal disorders) | 31 | 20 | 25 | 20
Dizziness (Nervous system disorders) | 24 | 26 | 25 | 25
Dyspepsia (Gastrointestinal disorders) | 13 | 25 | 13 | 16
Flushing (Vascular disorders) | 9 | 5 | 5 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 27 | 26 | 24 | 22
Oedema peripheral (General disorders) | 30 | 29 | 30 | 36
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 38 | 29 | 27
Weight decreased (Investigations) | 14 | 19 | 18 | 27
Diarrhoea (Gastrointestinal disorders) | 67 | 70 | 73 | 82
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 49 | 51 | 53 | 43
Night sweats (Skin and subcutaneous tissue disorders) | 7 | 10 | 12 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 16 | 19 | 17
Pericardial effusion (Cardiac disorders) | 3 | 9 | 10 | 7
Stomatitis (Gastrointestinal disorders) | 5 | 7 | 12 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 20 | 25 | 15 | 15
Bronchitis (Infections and infestations) | 14 | 5 | 16 | 11
Conjunctivitis (Infections and infestations) | 3 | 11 | 7 | 6
Decreased appetite (Metabolism and nutrition disorders) | 16 | 21 | 21 | 24
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 9 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 4 | 14 | 8
Vision blurred (Eye disorders) | 11 | 8 | 5 | 5
Vomiting (Gastrointestinal disorders) | 23 | 29 | 32 | 52
Abdominal distension (Gastrointestinal disorders) | 13 | 8 | 9 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 8 | 7 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 8 | 8 | 6
Gastritis (Gastrointestinal disorders) | 4 | 11 | 7 | 7
Headache (Nervous system disorders) | 75 | 73 | 60 | 76
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 13 | 15 | 18
Neutropenia (Blood and lymphatic system disorders) | 23 | 28 | 29 | 28
Pain (General disorders) | 19 | 10 | 12 | 10
Anxiety (Psychiatric disorders) | 6 | 9 | 15 | 12
Chills (General disorders) | 11 | 11 | 16 | 14
Depression (Psychiatric disorders) | 16 | 12 | 14 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 15 | 7 | 12
Flatulence (Gastrointestinal disorders) | 9 | 5 | 6 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 | 4 | 9 | 1
Influenza like illness (General disorders) | 14 | 17 | 9 | 13
Insomnia (Psychiatric disorders) | 19 | 20 | 14 | 12
Paraesthesia (Nervous system disorders) | 12 | 11 | 10 | 7
Periorbital oedema (Eye disorders) | 8 | 4 | 17 | 5
Pneumonia (Infections and infestations) | 5 | 5 | 10 | 13
Rash (Skin and subcutaneous tissue disorders) | 37 | 52 | 43 | 43
Toothache (Gastrointestinal disorders) | 10 | 15 | 8 | 8
Upper respiratory tract infection (Infections and infestations) | 28 | 26 | 35 | 23
Urinary tract infection (Infections and infestations) | 15 | 13 | 12 | 9
Weight increased (Investigations) | 18 | 8 | 13 | 11
Abdominal pain (Gastrointestinal disorders) | 25 | 26 | 24 | 20
Abdominal pain upper (Gastrointestinal disorders) | 13 | 24 | 17 | 18
Asthenia (General disorders) | 15 | 16 | 23 | 27
Contusion (Injury, poisoning and procedural complications) | 4 | 10 | 12 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 8 | 8 | 11
Influenza (Infections and infestations) | 13 | 4 | 17 | 11
Nausea (Gastrointestinal disorders) | 37 | 54 | 52 | 69
Neck pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 5 | 6
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 11 | 4 | 6
Pyrexia (General disorders) | 32 | 40 | 43 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.